CLINICAL TRIAL: NCT04686812
Title: Mexican Institute of Social Security and Companies' Collaboration Model to Promote Workers' Healthy Habits
Brief Title: Worksite Health Promotion Intervention to Promote Healthy Habits Among Workers From Mexican Companies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Collaborators: National Council of Science and Technology, Mexico (Other); University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Isabel Garcia-Rojas, Medical programs coordinator, Instituto Mexicano del Seguro Social
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SALUD-2005/02/14451
Record Dates: First submitted 2020-12-13; First posted 2020-12-29 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Cardiovascular Risk Factors
Keywords: workplace health promotion; intervention; Mexico

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Worksite health promotion program (Experimental): Participants had a baseline health risk assessment (HRA) after which they were invited to participate in a workplace health promotion program. The intervention lasted six months and included the following components: nutrition counseling, physical activity, and stress management. HRAs were performed 6 and 12 months after intervention onset.
  Interventions: Behavioral: Worksite health promotion program
- Control (No Intervention): Participants only had a baseline and follow-up health risk assessments at 6 and 12 months.

INTERVENTIONS:
Behavioral: Worksite health promotion program — Physical activity, nutrition, and stress management programs
  Other Names: Wellness intervention
  Arms: Worksite health promotion program

SUMMARY:
The purpose of this study is to explore the effects of a multidisciplinary worksite intervention program on biological cardiovascular risk factors.

DETAILED DESCRIPTION:
This prospective study consisted of a six-month company-based workplace health promotion intervention trial with a 6- and 12-month follow-up after the start of the intervention. IMSS' researchers promoted participation in this study among affiliated companies located in Mexico City and recruited 2,002 workers from seven different worksites, including a cooking utensils factory, a government public health services department, a metalworking company, a pharmaceutical company, a plastic factory, and a printing company. Companies were selected on the basis of their willingness to engage in the study's activities and consented to be part of either a control (n = 991, baseline and follow-up surveys only) or an intervention group (n = 1011, surveys plus intervention). Employers were presented with the intervention first and if they did not agree to participate, the option to enter the study as a control company was offered second. A health risk assessment (HRA), including a questionnaire and biological measurements (i.e., anthropometric and physiological measurements, as well as blood glucose, total cholesterol, triglycerides, and LDL), was performed at baseline, 6 months, and 1 year after the beginning of the study for both control and intervention groups.

IMSS researchers met in person with the directors of each company to introduce the intervention program and once they obtained authorization to perform the activities, nurses and social workers from the research team were in charge of promoting the intervention throughout the company. They held focus group meetings with workers during the workday, discussing the benefits of physical activity, healthy nutrition, and stress management. They also distributed flyers, displayed posters, and carried out one-on-one interactions whenever possible. As an incentive, they offered workers a complete and confidential physical examination, including blood work for free. They collected all data during the day shift and remained in each of the companies for about a week in order to enroll as many participants as possible but no further efforts were made to reach workers on sick leave or disability. Workers voluntarily participated.

Experts such as occupational physicians, nurses, psychologists, nutritionists, and sports medicine specialists designed the HRA questionnaire at IMSS. It included items on demographic and organizational characteristics, behavioral and biological risk factors for cardiovascular disease, and personal history of diabetes, hypertension, cardiovascular disease, and other self-reported medical conditions as doctors' diagnosis. The questionnaire was distributed among participating workers who completed it at home and submitted it to the research team on the day of their physical evaluation.

The physical examination included anthropometric (i.e., height, weight, waist circumference, and skinfold measurements to assess body fat, muscle, and bone mass), physiological measurements (such as heart rate, blood pressure, maximum oxygen intake), and a finger-stick cholesterol and glucose screening. These measurements and the survey information were used to determine the prevalence of individual cardiovascular risk factors (CVRF) such as age, income, gender, cardiorespiratory fitness, obesity, hypertension, diabetes, and dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

* Full-time employees of one of the participating companies
* Willing to participate in the baseline and follow-up health risk assessments and when applicable, in the different elements of the intervention.

Exclusion Criteria:

* Not being a full-time employee of the participating companies
* Refusing to participate in the health risk assessments and when applicable, in the different elements of the intervention

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2002 (Actual)
Dates: Start 2009-06-30 (Actual); Primary Completion 2011-06-30 (Actual); Study Completion 2011-06-30 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure from baseline to 6 and 12 months after a worksite health promotion intervention | Baseline, 6 months, and 12 months
  Blood pressure was measured manually by two research nurses using a sphygmomanometer and following protocols from the American Heart Association. Workers rested for about 5 minutes before the measurement, which was taken on their left arm while sitting.
Change in body mass index from baseline to 6 and 12 months after a worksite health promotion intervention | Baseline, 6 months, and 12 months
  Weight and height were measured in kg and cm, respectively, using a floor scale with stadiometer (Salter Brecknell brand). Workers were asked to remove their shoes and wore their usual clothing or uniform. Body mass index was calculated by dividing weight in kilograms by height in meters squared.
Change in oxygen uptake (VO2max) from baseline to 6 and 12 months after a worksite health promotion intervention | Baseline, 6 months, and 12 months
  The submaximum heart rate was obtained by applying Manero's protocol, which consisted on stepping up and down an ergometric bench. The frequency of each ascent was calculated as 90 for active workers and 84 for sedentary workers. One minute training was given to workers before the exercise to explain how to step up the bench (six steps to go up and six to come back down). The test lasted 5 minutes and was guided by an electronic metronome that marked the frequency of steps. A trained nurse measured each participant's heart rate by direct auscultation during the first 15 seconds immediately after the 5-minute exercise. This value was multiplied by 4 to obtain the sub-maximum heart rate and logged into a software that applied a correction factor by age and made group comparisons in Manero's nomograph, giving as a result the oxygen uptake in liters per minute.
Change in blood glucose levels from baseline to 6 and 12 months after a worksite health promotion intervention | Baseline, 6 months, and 12 months
  Levels of glucose were measured using a CardioChek® Plus analyzer (CCPA, PTS Diagnostics, model 2009). The materials used to take the test were alcohol swabs, sterile lancets, gloves, test strips, MEMo chip®, and the device CCPA.
Change in blood cholesterol levels from baseline to 6 and 12 months after a worksite health promotion intervention | Baseline, 6 months, and 12 months
  Levels of total cholesterol, LDL, and HDL were measured using a CardioChek® Plus analyzer (CCPA, People, Technology, and Service Diagnostics, model 2009). The materials used to take the test were alcohol swabs, sterile lancets, gloves, test strips, MEMo chip®, and the device CCPA.

CONTACTS AND LOCATIONS:
Overall Officials: Isabel J Garcia-Rojas, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Instituto Mexicano del Seguro Social, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
All data will be held in a public repository and Uniform Resource Locator (URL)/accession numbers will be available
Supporting Information: Study Protocol, ICF
Time Frame: The data will become available on January 31, 2021
Access Criteria: Information will be shared with peer-reviewers from journals where publications of this study will be submitted and with researchers needing information to include in review articles on the topics covered by this study. Requests for information will be reviewed by the principal investigator.
URL: http://fairsharing.org

REFERENCES:
- [Result] Garcia-Rojas IJ, Choi B, Krause N. Psychosocial job factors and biological cardiovascular risk factors in Mexican workers. Am J Ind Med. 2015 Mar;58(3):331-51. doi: 10.1002/ajim.22410. PMID 25678459
- [Result] Garcia Rojas, I. J. (2014). Associations of job strain, isostrain, and job insecurity with cardiovascular risk factors and productivity in Mexican workers. UCLA. ProQuest ID: GarciaRojas_ucla_0031D_10853. Merritt ID: ark:/13030/m5322105. Retrieved from https://escholarship.org/uc/item/2qd9m61x